CLINICAL TRIAL: NCT05554393
Title: A Measurable Residual Disease (MRD) Focused, Phase II Study of Venetoclax Plus Chemotherapy for Newly Diagnosed Younger Patients With Intermediate Risk Acute Myeloid Leukemia: A Tier 1 MYELOMATCH SubStudy
Brief Title: Comparing Cytarabine + Daunorubicin Therapy Versus Cytarabine + Daunorubicin + Venetoclax Versus Venetoclax + Azacitidine in Younger Patients With Intermediate Risk AML (A MyeloMATCH Treatment Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07534; NCI-2022-07534 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AL.6; MM1YA-CTG01 (Other: Canadian Cancer Trials Group); MM1YA-CTG01 (Other: CTEP); U10CA180863 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Specimen Handling; Cytarabine; Daunorubicin; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM I (daunorubicin, cytarabine, venetoclax) (Experimental): Patients receive daunorubicin IV on days 2-4, cytarabine IV continuously on days 2-8, and venetoclax PO QD on days 1-11. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of daunorubicin IV on days 2-3, cytarabine IV continuously on days 2-6, and venetoclax PO QD on days 1-8. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Venetoclax
- ARM II (azacitidine, venetoclax) (Experimental): Patients receive azacitidine IV or SC on days 1-7 or days 1-5 and 8-9 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for a total of 2 cycles, in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Drug: Azacitidine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Venetoclax
- ARM III (daunorubicin, cytarabine) (Active Comparator): Patients receive daunorubicin IV on days 1-3 and cytarabine IV, continuously, on days 1-7. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of cytarabine IV, continuously, on days 1-5 and daunorubicin IV on days 1-2. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacitidine; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
  Arms: ARM II (azacitidine, venetoclax)
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: ARM I (daunorubicin, cytarabine, venetoclax); ARM III (daunorubicin, cytarabine)
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
  Arms: ARM I (daunorubicin, cytarabine, venetoclax); ARM III (daunorubicin, cytarabine)
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: ARM I (daunorubicin, cytarabine, venetoclax); ARM II (azacitidine, venetoclax)

SUMMARY:
This phase II MyeloMATCH treatment trial compares cytarabine with daunorubicin versus cytarabine with daunorubicin and venetoclax versus venetoclax with azacitidine for the treatment of younger patients with intermediate risk acute myeloid leukemia (AML). Cytarabine is a drug that inhibits some of the enzymes needed for deoxyribonucleic acid (DNA) replication and repair and can slow or stop the growth of cancer cells. Daunorubicin is a drug that blocks a certain enzyme needed for cell division and DNA repair, and it may kill cancer cells. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Azacitidine is a drug that interacts with DNA to activate tumor-suppressing genes, resulting in an anti-tumor effect. Adding venetoclax to cytarabine and daunorubicin, and adding venetoclax to azacitidine, may work better than the usual treatment of cytarabine with daunorubicin alone. To decide if they are better, the study doctors are looking to see if venetoclax increases the rate of elimination of AML in participants by 20% or more compared to the usual approach.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the rates of undetectable measurable residual disease (MRD) in patients who achieve a complete remission (CR) after induction therapy with 7 +3 (cytarabine + daunorubicin hydrochloride [daunorubicin]) versus (vs.) azacitidine + venetoclax vs. 7+3 + venetoclax.

SECONDARY OBJECTIVES:

I. To estimate the frequency and severity of toxicities with each of the regimens.

II. To estimate complete remission (CR) rates (with and without MRD), complete remission with incomplete count recovery (CRi) (with and without MRD) rates, event-free survival (EFS), relapse-free survival (RFS), and overall survival (OS) with each of the regimens.

TERTIARY OBJECTIVES:

I. To evaluate response to therapy received according to genomic findings. II. To evaluate MRD kinetics by following patients with detectable MRD through Tier 2 and beyond.

III. To evaluate longer term outcomes by treatment arm, genomics, MRD outcome, and other features as patients receive additional myeloMATCH therapies to generate testable hypotheses for more precise patient selection for these therapies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive daunorubicin intravenously (IV) on days 2-4, cytarabine IV continuously on days 2-8, and venetoclax orally (PO) once per day (QD) on days 1-11. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of daunorubicin IV on days 2-3, cytarabine IV continuously on days 2-6, and venetoclax PO QD on days 1-8. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

ARM II: Patients receive azacitidine IV or subcutaneously (SC) on days 1-7 or days 1-5 and 8-9 and venetoclax PO on days 1-28 of each cycle. Cycles repeat every 28 days for a total of 2 cycles, in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

ARM III: Patients receive daunorubicin IV on days 1-3 and cytarabine IV, continuously, on days 1-7. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Based on a bone marrow aspiration assessment (completed at the discretion of the treating investigator), patients may receive reinduction consisting of cytarabine IV, continuously, on days 1-5 and daunorubicin IV on days 1-2. Cycle is 28 days and treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow aspiration and collection of blood samples on study and as clinically indicated.

After completion of study treatment, patients are followed up at 4 weeks, every 3 months for 1 year every 6 months for the second year and yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto MYELOMATCH and must have been given a treatment assignment to MyeloMATCH to MM1YA-CTG01 based on the presence of an actionable mutation as defined in MYELOMATCH
* Participants must have been registered to master screening and re-assessment protocol (myeloMATCH MSRP) prior to consenting to this study. Participants must have been assigned to this clinical trial, via MATCHBox Protocol Assignment Team, prior to registration to this study. Participants must have agreed to have specimens submitted for translational medicine (MRD) and must be offered the opportunity to submit biosamples for banking for future research as per the myeloMATCH MSRP

  * Note: Pre-enrollment/diagnosis labs must have already been performed under the MSRP
* Previously untreated, de novo acute myeloid leukemia (AML) defined by > 20% myeloblasts in the peripheral blood or bone marrow (refer to the 2016 updated World Health Organization [WHO] classification of myeloid neoplasms and acute leukemia) excluding all the following categories of AML:

  * Favorable cytogenetics: (t(8;21)q22;q22.1); RUNX1-RUNX1T1, inversion 16(p13.1;q22), t(16;16)(p13.1;q22); CBFB-MYH11
  * CEBPA biallelic mutations
  * NPM1 mutation
  * AML with PML-RARalpha
  * AML with any adverse cytogenetics, TP53 mutation, RUNX1 mutation, ASXL1, 11q23/KMT2 rearrangements
  * AML with FLT3-ITD or FLT3-TKD mutations
  * Therapy related AML, or AML following a diagnosis of myelodysplasia or myeloproliferative neoplasm Participants with central nervous system (CNS) disease are eligible for this trial and will be treated according to institutional guidelines with intrathecal chemotherapy for this aspect of their disease
* Age 18-59 years at time of induction therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) (must be done within 7 days of enrollment)
* Aspartate aminotransferase (AST) (serum glutamate pyruvate transaminase [SGPT]) +/or alanine aminotransferase (ALT) (serum glutamic-oxaloacetic transaminase [SGOT]) =< 3 × institutional ULN (must be done within 7 days of enrollment)
* Cardiac ejection fraction >= 50% (echocardiography or multigated acquisition scan [MUGA]) (if clinically indicated must be done within 14 days of enrollment)
* Calculated creatinine clearance >= 30 mL/min/ 1.73m^2; Clearance to be calculated using Cockcroft formula (must be done within 7 days of enrollment)
* White blood cells (WBC) must be < 25 x 10^9/L. Hydroxyurea and leukapheresis are permitted to control the WBC prior to enrollment and initiation of protocol-defined therapy but must be stopped at least 24 hours prior to the initiation of protocol therapy. 1 dose of cytarabine at 1 mg/m^2 for urgent cytoreduction is also permitted
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Males and females of reproductive potential must have agreed to use a highly effective contraceptive method while on treatment and for 6 months after stopping study drug. A woman is considered to be of "childbearing potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy/vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures.

Women of childbearing potential will have a pregnancy test to determine eligibility as part of the pre-study evaluation; this may include an ultrasound to rule-out pregnancy if a false-positive is suspected. Patient will be considered eligible if an ultrasound is negative for pregnancy

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Patients must be accessible for treatment, response assessment and follow up. Patients enrolled on this trial must be treated and followed at the participating centre. Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

Patients must agree to return to their primary care facility for any adverse events which may occur through the course of the trial

* In accordance with Canadian Cancer Trials Group (CCTG) policy, protocol treatment is to begin within 7 working days of patient enrollment
* Participants receiving strong or moderate CYP3A inhibitors must agree to discontinue use at least 48 hours prior to start of study treatment if assigned to arm 1 or 2
* Patients with known human immunodeficiency virus (HIV) infection who are on effective anti-retroviral therapy and have undetectable viral load within 6 months of enrollment are eligible for this trial
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load within 28 days of enrollment. Patients need to be on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection who have been treated and cured are eligible. Patients who with active HCV infection who are currently being treated must have an undetectable HCV viral load within 28 days of enrollment to be eligible

Exclusion Criteria:

* Prior therapy for AML except for hydroxyurea and leukapheresis to control blood counts. The use of all-trans retinoic acid (ATRA) is permitted until a diagnosis of acute promyelocytic leukemia, if suspected, is ruled out
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cytarabine, daunorubicin, azacitidine, venetoclax
* Pregnant women are excluded from this study because venetoclax, cytarabine and azacitidine have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with venetoclax, cytarabine and azacitidine breastfeeding should be discontinued if the mother is treated with venetoclax, cytarabine and azacitidine. These potential risks may also apply to other agents used in this study
* Patients with isolated myeloid sarcoma are not eligible
* Any other serious intercurrent illness, life threatening condition, organ system dysfunction, or medical condition judged by the local investigator to compromise the subject's safety (for example):

  * Active, uncontrolled bacterial, fungal, or viral infection

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurable residual disease (MRD) undetectable complete remission (CR) | Up to 2 cycles (56 days)
  Will assess after one induction cycle with or without the addition of venetoclax or two cycles of venetoclax and azacitidine. MRD by flow cytometry will be considered undetectable if ≤ 10^-3. The MRD negative CR will be assessed using European LeukemiaNet (ELN) 2017 criteria [Döhner 2017]. The analysis population for the primary outcome will be all randomized patients with the intent to treat population. The MRD undetectable CR rate will be the number of patients with MRD undetectable CR divided by the total number of patients. The differences of MRD undetectable CR rates between the experimental groups and the control group will be estimated and the corresponding one-sided 80% confidence limit will be calculated using Normal distribution approximation. MRD non-evaluable patients will be considered as MRD positive.

SECONDARY OUTCOMES:
Frequency and severity of toxicities with each of the regimens | Up to 10 years
  All patients who have received at least one dose of study treatment will be included in the safety analysis. Adverse events will be graded using the Common Terminology Criteria for Adverse Events version 5.0. The incidence of adverse events will be summarized by type severity and relationship to the study drugs. A Fisher's exact test will be used to compare toxicities between the two arms, if needed.
CR rates | Up to 2 cycles (56 days)
  Will be assessed per 2017 ELN guidelines and will be tabulated. Exact 95% confidence intervals will be calculated.
Complete remission with incomplete count recovery (CRi) | Up to 2 cycles (56 days)
  Will be assessed with and without MRD. Will be assessed per 2017 ELN guidelines and will be tabulated. Exact 95% confidence intervals will be calculated.
Event-free survival | From the date of randomization to the first: date of primary refractory disease; date of progressive disease; date off protocol therapy without CR or CRi; date of relapse from CR or CRi, or death from any cause, assessed up to 10 years
  Patients not known to have any of these events are censored on the date of last contact. Will be described by the Kaplan-Meier estimate, and log-rank tests will be used to test the difference between each experimental arms to the control arms.
Relapse-free survival | From the time of CR or CRi, until the relapse from CR or CRi, or death from any cause, assessed up to 10 years
  Will be calculated for participants who have achieved a CR or CRi. For patients who have not relapsed or died, will be censored on the date of the last disease assessment. Will be described by the Kaplan-Meier estimate, and log-rank tests will be used to test the difference between each experimental arms to the control arms.
Overall survival | From randomization to the time of death from any cause, assessed up to 10 years
  For patients who did not die, overall survival time will be censored at the time of last known alive date. Will be described by the Kaplan-Meier estimate, and log-rank tests will be used to test the difference between each experimental arms to the control arms.
Responses to therapy received relative to genomic findings | Up to 10 years
  Will evaluate to gain insights toward more precise patient selection for optimal outcomes.

OTHER OUTCOMES:
Comparative analysis by molecular characteristics | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary L Savoie, Principal Investigator — Canadian Cancer Trials Group
Locations (171):
- United States (161):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Memorial Hospital West, Pembroke Pines, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (8):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm